CLINICAL TRIAL: NCT04010201
Title: A Registered Cohort Study on Brain Calcification
Status: Recruiting | Type: Observational
Sponsor: Wan-Jin Chen (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor-Investigator, Wan-Jin Chen, The Vice-Director for the Department of Neurology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2019]198
Record Dates: First submitted 2019-07-04; First posted 2019-07-08 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Brain Calcification
Keywords: brain calcification; natural history; genetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brain calcification is a common neuroimaging feature in patients with metabolic, neurological, or developmental disorders, infectious diseases, traumatic or toxic history, as well as in otherwise normal older people. To understand the clinical and genetic characteristics of brain calcification, we establish a cohort of brain calcification to follow up patients with brain calcification.

ELIGIBILITY:
Inclusion Criteria:

* Patients with brain calcium deposit(s) based on examinations of CT scans
* Patients with total calcification score(TCS) greater than the physiological threshold
* Relatives of brain calcification patients.
* Unrelated healthy controls
* Participants or Parent(s)/legal guardian(s) willing and able to complete the informed consent process

Exclusion Criteria:

* Brain calcification caused by specific secondary factors such as infection, poisoning, and trauma
* Participants declining or unable to comply with trial procedures and visit schedule

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Brain calcification patients who are diagnosed in the First Affiliated Hospital of Fujian Medical University
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-08-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2079-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hereditary brain calcification | Up to 20 years
  Look for the causative gene in the patient with brian calcification

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No